CLINICAL TRIAL: NCT02583399
Title: A Multi-Center, Open-Label Pharmacokinetic and Safety Study for Reduction in Fever or Management of Pain in Pediatric Subjects Aged Birth to Six Months
Brief Title: Safety and Pharmacokinetic Study of Intravenous Ibuprofen in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL-022
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Pain; Fever
Keywords: Pediatric (Birth to less than 6 months of age); Pain; Fever
MeSH Terms: conditions — Pain; Fever | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Multi-center, Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibuprofen (Experimental): Ibuprofen, 10 mg/kg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen, 10 mg/kg

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic profile of a single dose of intravenous ibuprofen administered over approximately ten (10) minutes.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the pharmacokinetic profile of a single dose of intravenous ibuprofen administered over approximately ten (10) minutes.

ELIGIBILITY:
Inclusion Criteria:

* Be a hospitalized male or female subject between birth (> 37 weeks gestational age) and < six (6) months of age.
* Have a clinical indication of pain or fever.
* Have written informed consent provided by legal parent, guardian, or authorized agent prior to participation in the study or performance of any study-only related procedures.

Exclusion Criteria:

* Have inadequate intravenous access.
* Have an uncorrected ductus dependent congenital heart disease.
* Have any history of allergy or hypersensitivity to non-steroidal anti-inflammatory drug or aspirin.
* Have a current history of uncorrected hypovolemia or acute renal disease.
* Have a current history of acute liver disease.
* Have received NSAID, acetaminophen, or aspirin drug therapy within four hours prior to dosing. Have received another investigational drug within the past 30 days.
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rice, MD, Study Chair — Vanderbilt University
Locations (4):
- United States (4):
  - Kosair Charaties Pediatric Research Unit, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glover CD, Berkenbosch JW, Taylor MB, Patel NV, Kaelin B, Gibson BHY, Zhong J. A Multi-Center Evaluation of the Pharmacokinetics and Safety of Intravenous Ibuprofen in Infants 1-6 Months of Age. Paediatr Drugs. 2023 Sep;25(5):585-593. doi: 10.1007/s40272-023-00576-9. Epub 2023 Jun 9. PMID 37294477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between 08-Aug2017 and 21-Feb2019. Subject were recruited were hospitalized pediatric subjects, aged birth (greater than 37 weeks gestational age) to less than six months of age, with a clinical indication of pain and fever.
Period: Overall Study
Arm/Group | Ibuprofen
Started | 30
Completed | 24
Not Completed | 6
Not completed — Able to be discharged | 3
Not completed — Wanted to use a restricted medication | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ibuprofen
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: days] | 127.7 (33.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  White | 17
  Other | 4
  Hispanic/Latino | 5
  Non-Hispanic/Non-Latino | 19
Weight [Mean (Standard Deviation); unit: kilograms] | 6 (1.45)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) 0-4 Hours of a Single Dose of Intravenous Ibuprofen (IVIb) Administered Over 5-7 Minutes.
Description: This outcome measurement was to the determine the area under the plot of plasma concentrations of drug against time after drug administration. Pharmacokinetic samples were collected immediately following the first dose, the utilizing sparse sampling techniques, samples were collected at 30 minutes, 1 hour, 2 hours and 4 hours.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: mcg*hr/mL
Arm/Group | Ibuprofen
Number analyzed (Participants) | 24
mcg*hr/mL | 75.74 (4.09)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of a Single Dose of Intravenous Ibuprofen (IVIb) Administered Over 5-7 Minutes.
Description: This outcome measurement was to measure the maximal or peak measured serum concentration (Cmax) of a single dose of intravenous ibuprofen (IVIb) after its administration. Pharmacokinetic samples were collected immediately following the first dose, the utilizing sparse sampling techniques, samples were collected at 30 minutes, 1 hour, 2 hours and 4 hours.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: microgram/milliliter
Arm/Group | Ibuprofen
Number analyzed (Participants) | 24
microgram/milliliter | 56.28 (2.77)

3. Primary Outcome: Elimination Half Life (T 1/2) of a Single Dose of Intravenous Ibuprofen (IVIb) Administered Over 5-7 Minutes.
Description: This outcome measurement was to determine the half-life or the period of time required for the concentration or amount of drug in the body to be reduced to exactly one-half of a given concentration or amount. Pharmacokinetic samples were collected immediately following the first dose, the utilizing sparse sampling techniques, samples were collected at 30 minutes, 1 hour, 2 hours and 4 hours.
Time Frame: 4 hours
Population: Analysis were performed using sparse sampling concentration. Phoenix WinNonlin treats the sparse data as a special case of plasma concentration data. The NCA sparse methodology calculates PK parameters based on the mean profile for all the subjects in the dataset. Consequently, standard deviation can only be calculated based on observed data (AUC0-t and Cmax) but not on derived data (Tmax, T½ el.)
Measure: Number; unit: hours
Arm/Group | Ibuprofen
Number analyzed (Participants) | 24
hours | 1.30

4. Primary Outcome: Time to Maximum Concentration (Tmax) of a Single Dose of Intravenous Ibuprofen (IVIb) Administered Over 5-7 Minutes.
Description: This outcome measurement was to determine the time to maximum concentration (Tmax) of a single dose of intravenous ibuprofen (IVIb) after its administration. Pharmacokinetic samples were collected immediately following the first dose, the utilizing sparse sampling techniques, samples were collected at 30 minutes, 1 hour, 2 hours and 4 hours.
Time Frame: 4 hours
Population: as for outcome 3
Measure: Number; unit: minutes
Arm/Group | Ibuprofen
Number analyzed (Participants) | 24
minutes | 10

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the treatment period beginning with the start of the study drug administration through study hour 72 or until discharge, whichever occurs first.
Arm/Group | Ibuprofen
All-Cause Mortality (participants affected / at risk) | 8/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=24)
Pericardial effusion (Cardiac disorders) | 1 (1)
Chylothorax (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=24)
Eye discharge (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Post-procedural fever (Injury, poisoning and procedural complications) | 1 (1)
White blood cells increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripherial artery thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT02583399/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT02583399/SAP_001.pdf